CLINICAL TRIAL: NCT06393764
Title: Establishment of a Patient-based Cohort : Cancer-related Venous Thromboembolic Disease.
Brief Title: Cancer-related Venous Thromboembolic Disease - Cohort Study
Acronym: CAPE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0290
Record Dates: First submitted 2024-04-19; First posted 2024-05-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Thrombosis Embolism; Thromboses, Venous; Cancer
MeSH Terms: conditions — Embolism and Thrombosis; Venous Thrombosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collected at inclusion (66.4 ml) and in case of recurrence of thrombo-embolic venous disease ( 54.5 mL) to store plasma, serum, DNA and RNA.t Tumor tissue collection (taken during excision or biopsy as part of routine care) Urine (20 to 40 mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer patients treated for MVTE: All the patients are included in one arm. They will undergo various type of samples.
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — Collecte of blood and urine samples

SUMMARY:
Venous thromboembolic disease (VTE) is a common (1/1000), potentially serious disease (10% mortality when the clinical presentation is that of pulmonary embolism (PE)). In cancer patients, the risk of developing VTE is high and constitutes a negative prognostic factor for cancer; the risk of bleeding is also increased. The study of VTE in the context of cancer is a major challenge, given the frequency of the association, the heterogeneity of the situations, the risk factors involved and the therapeutic issues in both curative and primary prevention; in this field, many uncertainties remain, justifying a study focused on the association of VTE and cancer.

DETAILED DESCRIPTION:
Cancer is associated with a higher risk of VTE and mortality. This association is characterized by various uncertainties at pathophysiological, diagnostic, therapeutic and prognostic levels.

CAPE STUDY is a prospective, single-center interventional cohort follow-up study designed to investigate the risk of recurrence of VTE and its mechanisms in cancer patients.

The study involves the collection of biological samples from cancer patients with venous thromboembolic disease.

At inclusion and in case of recurrence of thrombosis or hemorrhage:

* Blood samples will be taken for analysis and to constitute a biobank for future assays.
* Urine samples will be collected Once a year for 5 years (and adapted to the clinical context): visit as part of routine care, or mailing of a questionnaire, or telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and more.
* Patients with active cancer or requiring cancer treatment at the time of their VTE episode
* Patients with documented VTE less than 2 years old
* Patients affiliated to the social security system
* Patient who has signed a written informed consent

Exclusion Criteria:

* Patient under 18
* Refusal to participate
* Incapacity to consent to the study
* Patient under guardianship
* Incapacity to communicate (comprehension disorder)
* Life expectancy of less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major cancer patients with venous thromboembolic disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2034-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolic recurrence | 5 years
  Venous thromboembolic recurrence

SECONDARY OUTCOMES:
Major hemorrhage | As long as the patient is on anticoagulant treatment during the 5 years of follow-up
  Fatal haemorrhage, clinical haemorrhage associated with a fall in haemoglobin of 2g/dl or more, clear clinical haemorrhage requiring transfusion of at least 2 red blood cells packed, intracranial, medullary, retroperitoneal, pericardial, intra-articular, intra-muscular, intra-ocular, intra-pulmonary haemorrhage, any other haemorrhage considered serious by the investigator
Mortality | 5 years
  Global (all causes) and secondary to recurrent VTE or hemorrhage
Arterial events | 5 years
  Atrial fibrillation, cerebrovascular accident, coronary accident, arteriopathy of the lower limbs, digestive vascular accident (splanchnic, renal, mesenteric etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Françis Couturaud, Pr, Principal Investigator — CHU Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement